CLINICAL TRIAL: NCT02807155
Title: Helmsley Type 1 Diabetes Youth Transitional Program
Brief Title: Let's Empower and Prepare Young Adults With Type 1 Diabetes
Acronym: LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Anne Peters, Professor of Clinical Medicine, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010PG-T1D011
Record Dates: First submitted 2016-06-15; First posted 2016-06-21 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Transitional Care; Young Adult; Guided Imagery
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — tetraethylpyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non-Intervention Control (No Intervention): No intervention will be delivered.
- Continuity Group (Experimental): Continuity Group participants aged 20-21 (i.e. the last year of the LEAP Program) will be seen at one of the 2 study centers - 1) the newly established LAC+USC Diabetes Transition Clinic; or 2) Children's Hospital Los Angeles Pediatric Endocrinology Clinic, and will receive the full 1-year Transition Empowerment Program - Continuity Group"
  Interventions: Behavioral: Transition Empowerment Program; Behavioral: Transition Empowerment Program (TEP) + Diabetes Wellness Council (DWC)
- Rescue Group (Experimental): Rescue Group participants aged 21-25 will be connected to a diabetes healthcare "home" (medical clinic or doctor's office) in Los Angeles County based on geography and personal preference. Those individuals connected to the LAC+USC Diabetes Transition Clinic will receive the full 1-year Transition Empowerment Program - Rescue Group" (TEP-RG). Those assigned to other providers in LA County will have access to the web-based curriculum.
  Interventions: Behavioral: Online Transition Empowement Program Access

INTERVENTIONS:
Behavioral: Transition Empowerment Program — Participants will receive the 1-year transition empowerment program/curriculum (TEP-CG) alone.
  Other Names: TEP
  Arms: Continuity Group
Behavioral: Transition Empowerment Program (TEP) + Diabetes Wellness Council (DWC) — Participants will receive the identical 1-year Transition Empowerment Program, plus the innovative wellness-based group process (council).
  Other Names: TEP + DWP
  Arms: Continuity Group
Behavioral: Online Transition Empowement Program Access — Participants assigned to an outside medical home would be followed according to the clinical needs as assessed by their medical provider. They would be given access to the TEP website curriculum, but would not participate in other aspects of the 1-year TEP.
  Arms: Rescue Group

SUMMARY:
In Los Angeles County, the most populous county in the United States, there are an estimated 8,000 children under the age of 21 with type 1 diabetes. Although provisions for pediatric care exist, once these children become young adults they age out of their health care services. There is no formal transitional care program to help these individuals through this process of changing health plans and many end up without adequate care. This project aims to develop and implement a transition care program for young adults with type 1 diabetes in order to ensure uninterrupted transition from pediatric to adult diabetes health care and improve health and psychological outcomes.

DETAILED DESCRIPTION:
The Final LEAP Program is a one year curriculum designed to give young adults with type 1 diabetes the skills to effectively transfer from pediatric to adult care without lapse in medical treatment. The Final LEAP curriculum consists of four modules; 1) back-to-basics diabetes education, 2) handling daily life with diabetes, 3) navigating the healthcare system/transitioning, and 4) issues relating to sex, drugs and alcohol. Additionally, the program includes quarterly group classes covering topics such as enrolling into a Los Angeles County Health Care Plan, carbohydrate counting, and community connections. Each individual module will be introduced in packet form 3 months before the scheduled clinic appointments. At each clinic appointment throughout the year the modules will be taught and a post-test will be given to assess knowledge. Study participants will continue their standard diabetes clinic appointments, which occur every 3 months. At these visits, the study team will collect an additional HbA1C at baseline, 6mo, and 12mo of the correlating study/standard visit. An HbA1c test will be performed during their standard diabetes clinic appointment using the "DCA 2000", which requires an additional patient-administered finger stick. Protected Health Information will be accessed through medical records for those participants consented into the Continuity Control and Intervention groups. Measures gathered at baseline, 6 months, and 12 months will be height, weight, BMI, lipid panel, and insulin regiment. Apart from the DCA 2000 HbA1c measurement, all three clinics assess HbA1c using a laboratory and these results are recorded in the patient's chart. HbA1c obtained through lab measurements will be abstracted from the patients chart at baseline, 3 months, 6 months, 9 months, and 12 months.Additionally, 25 participants will be selected to take part in an empowerment group as part of the intervention. The participants will be chosen at random. The empowerment group will meet monthly, either in the evening or on a weekend. 10 -12 participants will gather and will have the opportunity to talk about issues affecting their lives in regards to diabetes. . We are looking to see if participation in an empowerment group has positive results on a person's diabetes care.Rescue Group - Participants will be assigned to either the Los Angeles County + University of Southern California (LAC+USC) Diabetes Transition Clinic (Experimental Group) or to a clinic near their home, based on their choice.Continuity Group - The Continuity Intervention Group will be recruited from among current patients attending the pediatric diabetes clinics at the 2 study sites, LAC+USC and Children's Hospital Los Angeles (CHLA) and assigned to the experimental group. Participants will receive the 1-year Final LEAP program. Half of the participants will be randomized to participate in the Diabetes Wellness Council and these results will be compared to those who did not participate. The Continuity control group will be individuals followed at Children's Hospital Orange County (CHOC) receiving standard care. The control group participants will meet the same inclusion/exclusion criteria as those in the experimental group.STATISTICS: For the Rescue group, 100 participants in each group would be sufficient to detect an effect of .4, a moderate effect, which translates into a difference in change of A1C of .49%. For the Continuity group, at the proposed sample sizes of 50-50-100, it would be possible to detect a difference for an omnibus ANOVA of an effect size of .22, a small effect. This would translate into a difference across groups in change of A1C of .27%.PLANS FOR ANALYSIS: Both experimental and control group participants will assessed at 6 and 12 months for A1c and psychosocial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 25 at time of enrollment
* Diagnosis of type 1 diabetes according to American Diabetes Association for at least two years
* Receiving routine diabetes care by an assigned provider
* in the last year of pediatric care (defined as anticipating transition to adult care within the next year)

Exclusion Criteria:

* Pregnant or planning to become pregnant within 12 months

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Number of Routine Diabetes Clinic Visits | 12 Months

SECONDARY OUTCOMES:
Hemoglobin A1C | 12 Months
Incidence of Hypoglycemia | 12 Months
Health Care Utilization | 12 Months
Diabetes Empowerment Scale- Short Form | 12 Months
Diabetes Knowledge Test- Adapted | 12 Months
Perceived Stress Scale- Adapted | 12 Months
Patient Health Questionnaire-9 | 12 Months
Satisfaction with Life Scale | 12 Months
Arizona Integrative Outcomes Scale | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Anne L Peters, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weigensberg MJ, Vigen C, Sequeira P, Spruijt-Metz D, Juarez M, Florindez D, Provisor J, Peters A, Pyatak EA. Diabetes Empowerment Council: Integrative Pilot Intervention for Transitioning Young Adults With Type 1 Diabetes. Glob Adv Health Med. 2018 Mar 8;7:2164956118761808. doi: 10.1177/2164956118761808. eCollection 2018. PMID 29552422